CLINICAL TRIAL: NCT00112229
Title: Immunotherapy of HLA-A2 Positive Stage III/IV Melanoma Patients With CpG7909, Tumor Antigenic Peptides and Montanide
Brief Title: Immunotherapy of HLA-A2 Positive Stage III/IV Melanoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Ludwig Institute for Cancer Research (Other)
Responsible Party: Principal Investigator, Prof Olivier Michielin, M.D., Ph.D., Professor, Centre Hospitalier Universitaire Vaudois
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUD 2000-018
Record Dates: First submitted 2005-05-31; First posted 2005-06-01 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Melanoma
Keywords: Immunotherapy; Vaccination; Melanoma; Melan-A/Mart-1 peptide; Tyrosinase peptide; CpG; Montanide
MeSH Terms: conditions — Melanoma

ARMS (4):
- group 1 (Experimental): Melan-A analog peptide + CpG + Montanide
  Interventions: Biological: group 1
- group 2 (Experimental): Melan-A natural peptide + CpG + Montanide
  Interventions: Biological: group 2
- group 3 (Experimental): Melan-A natural peptide + Tyrosinase YMD peptide + CpG + Montanide
  Interventions: Biological: group 3
- group 4 (Experimental): Melan-A analog peptide + Tyrosinase YMD peptide + CpG + Montanide
  Interventions: Biological: group 4

INTERVENTIONS:
Biological: group 1 — Melan-A analog peptide + CpG + Montanide
  Arms: group 1
Biological: group 2 — Melan-A natural peptide + CpG + Montanide
  Arms: group 2
Biological: group 3 — Melan-A natural peptide + Tyrosinase YMD peptide + CpG + Montanide
  Arms: group 3
Biological: group 4 — Melan-A analog peptide + Tyrosinase YMD peptide + CpG + Montanide
  Arms: group 4

SUMMARY:
The purpose of this study is to determine whether vaccination with tumor antigenic peptides and both CpG and Montanide adjuvants can induce an immune response in melanoma patients and to assess the safety of this vaccination.

DETAILED DESCRIPTION:
Immune therapy with tumor antigenic peptides is generally quite well tolerated. However, immune activation is often only weak or even undetectable, and clinical responses (supposedly corresponding to protective immunity) are unfortunately infrequent. Further progress is required to improve the vaccines, with the goal to increase the strength of immune activation.

The tumor antigenic peptides Melan-A/Mart-1 (EAA and ELA) and Tyrosinase (YMD) are combined with two drugs in this study, both of which are known to enhance immune responses: first, CpG 7909 oligodeoxynucleotides, and second, Montanide ISA-51.

* Group 1: vaccination with Melan-A analog peptide + CpG and Montanide adjuvants;
* Group 2: vaccination with Melan-A natural peptide + CpG and Montanide adjuvants;
* Group 3 : vaccination with Melan-A natural and Tyrosinase peptides + CpG and Montanide adjuvants;
* Group 4 : vaccination with Melan-A analog and Tyrosinase peptides + CpG and Montanide adjuvants.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage III or stage IV melanoma
* Tumor expression of Melan-A +/- Tyrosinase
* Human leukocyte antigen-A2 (HLA-A2) positive

Exclusion Criteria:

* Clinically significant heart disease
* Serious illnesses, eg, serious infections requiring antibiotics, bleeding disorders or uncontrolled peptic ulcer, or seizure or central nervous system disorders
* History of immunodeficiency disease or autoimmune disease
* Coagulation or bleeding disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2003-04; Primary Completion 2011-08 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Melan-A and Tyrosinase specific CD8+ T-cell reactivity will be measured by Tetramers and Elispot assays | Change from baseline in CD8 T-cells reactivity at day 375
Safety of vaccination will be assessed according to National Cancer Institute Common Toxicity Criteria (NCI CTC) scale | Change from baseline to day 375

SECONDARY OUTCOMES:
In patients with measurable disease, tumor response will be assessed radiologically | Change from baseline in tumor response at day 375

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Michielin, MD, Principal Investigator — Ludwig Institute for Cancer Research
Locations (1):
- Ludwig Institute for Cancer Research + Multidisciplinary Oncology Center at the Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Result] Speiser DE, Lienard D, Rufer N, Rubio-Godoy V, Rimoldi D, Lejeune F, Krieg AM, Cerottini JC, Romero P. Rapid and strong human CD8+ T cell responses to vaccination with peptide, IFA, and CpG oligodeoxynucleotide 7909. J Clin Invest. 2005 Mar;115(3):739-46. doi: 10.1172/JCI23373. PMID 15696196
- [Result] Baumgaertner P, Jandus C, Rivals JP, Derre L, Lovgren T, Baitsch L, Guillaume P, Luescher IF, Berthod G, Matter M, Rufer N, Michielin O, Speiser DE. Vaccination-induced functional competence of circulating human tumor-specific CD8 T-cells. Int J Cancer. 2012 Jun 1;130(11):2607-17. doi: 10.1002/ijc.26297. Epub 2011 Aug 24. PMID 21796616